CLINICAL TRIAL: NCT03731143
Title: A Simple Surgical Approach for the Management of Acquired Severe Lower Punctual Stenosis
Brief Title: Management of Lower Punctal Stenosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Sameh S. Mandour, Assistant Professor of Ophthalmology., Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 446H/2013
Record Dates: First submitted 2018-10-26; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Epiphora
Keywords: pigtail; punctal stenosis; bicanalicular
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): surgical opening the lower punctum using the pig tail probe and a scalpel followed by insertion of self retaining bicanalicular stent (FCI®; Paris, France).
  Interventions: Procedure: insertion of self retaining bicanalicular stent

INTERVENTIONS:
Procedure: insertion of self retaining bicanalicular stent — The pigtail probe was passed through the canalicular system from the normal punctum to the occluded aspect. When the tip of the pigtail probe was positioned near the occluded punctal area, the surgeon pushed the area to be tented with the pigtail probe. After they advanced the pigtail probe back and forth several times until they could locate the correct position of the occluded punctum, the authors incised the tented area with a scalpel No. 11 to make a new punctal opening.
  To ensure punctal and canalicular patency, syringing was repeated through the perforated punctum. To prevent re-occlusion of punctal opening, a self retaining bicanalicular tube (FCI®; Paris, France) was inserted through the normal and perforated puncti

SUMMARY:
a prospective non-randomized study conducted upon 24 patients with severe lower punctual stenosis (grade 0 according to Kashkouli scale) attending at Menoufia University hospitals. The upper punctum and canaliculus were patent. All patients were complaining of epiphora and had a thorough ophthalmological examination including dye disappearance test, and slit-lamp examination. Pigtail probe was used from patent upper punctum to detect the lower stenosed punctum which was opened with a scalpel. Syringing of the lower lacrimal passages was done to confirm its patency and self retaining silicone bicanalicular stent was inserted. The silicone tube was left in place for 6 months before it was removed. Patients were then followed up for 1 year after the surgery.

DETAILED DESCRIPTION:
This is a prospective non-randomized study which was conducted upon 24 patients with total lower punctual occlusion attending at Menoufia University hospitals in the period from January 2014 to January 2018. Ethics approval from the institutional review board was obtained, and a written informed consent was taken from every patient according to the Declaration of Helsinki.

All patients of the study were complaining of epiphora and had a thorough ophthalmological examination including dye disappearance test, and slit-lamp examination. The dye disappearance test was performed with a drop of 2% fluorescein sodium and assessment after 5 minutes of the remaining dye in the tear meniscus was done and results were graded.

Surgical procedure

All operations were done under general anesthesia and were performed by two authors (SSM, KES). The authors performed lacrimal probing and syringing test through the normal punctum to exclude concomitant occluded common canaliculus or nasolacrimal duct. The pigtail probe was passed through the canalicular system from the normal punctum to the occluded aspect. When the tip of the pigtail probe was positioned near the occluded punctal area, the surgeon pushed the area to be tented with the pigtail probe. After they advanced the pigtail probe back and forth several times until they could locate the correct position of the occluded punctum, the authors incised the tented area with a scalpel No. 11 to make a new punctal opening.

To ensure punctal and canalicular patency, syringing was repeated through the perforated punctum. To prevent re-occlusion of punctal opening, a self retaining bicanalicular tube (FCI®; Paris, France) was inserted through the normal and perforated puncti.

The silicone tube was left in place for 6 months before it was removed. Patients were then followed up for 1 year after the surgery (6 months after removal of the tube). During the follow-up period, the authors investigated the improvement of subjective epiphora symptoms based on Munk score, fluorescein disappearance test, maintenance of newly formed punctal opening, and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

1. severe lowee punctual stenosis
2. patent upper punctum and canaliculus as well as patent nasolacrimal duct
3. normal lower eyelid margin position -

Exclusion Criteria:

1. patients with punctal stenosis with grades more than 0 according to Kashkouli scale
2. patients with previous eyelid surgery
3. a lump overlying or involving the punctum or other part of the tear drainage system.

Ages: 17 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-12 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Degree of improvement of epiphora by Munk score | 1 year
  Measurement of improvement of epiphora by use of Munk score as follow Grade Clinical finding 0 No Epiphora.
  1. Occasional epiphora requiring drying or dabbing less than twice a day.
  2. Epiphora requiring dabbing two to four times per day.
  3. Epiphora requiring dabbing five to ten times per day.
  4. Epiphora requiring dabbing more than ten times daily or constant tearing.
Degree of improvement of lacrimal drainage by Dye disappearance test | 1 year
  measurement of improvement by using the dye disappearance test. It was performed by putting a drop of 2% fluorescein sodium in the conjunctival sac followed by assessment after 5 minutes of the remaining dye in the tear meniscus. Results were graded according to the following scale
  Grade Dye disappearance time, min
  1. <3
  2. 3-5
  3. >5
Slit lamp assesment of the state of the lower punctum | 1 year
  Slit lamp examination of the lower punctum and its grading according to Kashkouli scale as follows:
  Grade Clinical Findings 0 No punctum (agenesis)
  1. Papilla is covered with a membrane (difficult to recognize)
  2. Less than normal size, but recognizable
  3. Normal
  4. Small slit (<2 mm)
  5. Large slit (≤2 mm

CONTACTS AND LOCATIONS:
Overall Officials: Sameh S Mandour, MD, Principal Investigator — Menoufia Fculty of Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mandour SS, Said-Ahmed KE, Khairy HA, Elsawy MF, Zaky MA. A Simple Surgical Approach for the Management of Acquired Severe Lower Punctal Stenosis. J Ophthalmol. 2019 Jan 14;2019:3561857. doi: 10.1155/2019/3561857. eCollection 2019. PMID 30733874